CLINICAL TRIAL: NCT05130164
Title: Forensic Assessment of Age From Pulp Cavity Using Cone Beam Computed Tomographic Images (An Observational Cross- Sectional Study)
Brief Title: Age Estimation From Pulp Cavity Analysis Using Cone Beam Computed Tomographic Images for Forensic Purposes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Christine Atef Banoub Beshara, Principal investigator & PhD student, Cairo University
Other Study IDs: Christine Atef ORAD 7-1-1
Record Dates: First submitted 2021-11-08; First posted 2021-11-22 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Healthy
Keywords: CBCT; Forensic dentistry; Age determination by teeth

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single group: Single group will be selected for age estimation using CBCT Scans
  Interventions: Radiation: CBCT

INTERVENTIONS:
Radiation: CBCT — Cone beam computed tomographic images selected for age estimation

SUMMARY:
Forensic odontology is a branch of forensic science that utilizes a dentist's expertise in identification of individuals for whom traditional methods of identification aren't accessible due to a lack of common identification features. Medico-legal issues, natural catastrophes such as tsunamis, earthquakes, and explosions, death verification in monetary concerns, religious and social reasons are all examples of situations that require identification. Age, stature, sex and ethnicity are the "big four" determinants of personal identification. Dental age estimation has the benefit of that teeth are less influenced by external physical, chemical, or mechanical variables than other portions of the skeleton. Secondary dentin deposition in human teeth progresses with age that results in reduction in the size of the tooth pulp cavity which can be assessed as an age indicator. A significant relationship between pulp width and age was originally discovered in a study by Kvaal et al., 1995 who created regression formulae for age prediction using periapical radiograph by measuring of pulp size. Also, the assessment of pulp/tooth volume ratio relying on the gradual reduction in pulp volume produced by continuous apposition of dentin during life is one well-known dental age estimation approach. Cone beam computed tomography (CBCT) provides accurate three-dimensional images of the maxillofacial area. In addition, CBCT may be beneficial in some forensic situations, as it has massive benefits for post-mortem forensic imaging, as it offers skeletal imaging with high resolution, cheap cost, simplicity and portability. CBCT can be used in forensic age assessment since it is non-invasive and allows for the reconstruction of images in multiple planes to display anatomical and imaged elements in distinct planes. Our hypothesis is that pulp space analysis is totally different between different ages and that there is a correlation between age and pulp space analysis that could be of a forensic significance for age estimation in the investigated population.

DETAILED DESCRIPTION:
In this observational cross-sectional study, cone beam computed tomography scans will be recruited that are with the required complement of teeth and in the age range between 20 and 60 years then, correlation between chronological age versus cone beam computed tomography age through pulp space analysis will be done by two methods which are linear measurements and volumetric measurements of pulp and tooth size. First, linear measurements will be done according to kvaal's et al approach, measurements from mandibular lateral incisors, canines and first premolars and maxillary central and lateral incisors and second premolars were most strongly correlated with age, so these teeth will be selected for the investigation. A paired t-test on these measurements showed that there were no significant differences between teeth from the left and the right side of the jaw. Consequently, teeth from either the left or the right side will be chosen, whichever will be best suited for measurement. Not knowing the age and gender of the individual, the following measurements will be carried out on the radiographs of all six types of teeth: the maximum tooth length (T), pulp length and root length (R) on the mesial surface from the enamel-cementum junction (ECJ) to the root apex, the root and pulp width both at the ECJ (level A) and at the midroot level, i.e. halfway between the ECJ and the apex of the root (level C), as well as at the midpoint between the ECJ and midroot level (level B). Second, volumetric Measurements will be done to calculate pulp/ tooth volume ratio.

ELIGIBILITY:
Inclusion Criteria:

* CBCT scans for male and female Egyptians between the ages of 20 and 60 years.
* CBCT scans with the required complement of teeth.

Exclusion Criteria:

* CBCT scans that lack a proof of age or date of birth.
* CBCT scans with the required teeth showing pathological processes in the apical bone.
* CBCT scans with overlying teeth.
* CBCT scans in which the required teeth were filled, prosthetically restored or carious.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: CBCT scans that meet the eligibility criteria for age estimation
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2022-04-02 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Pulp/ tooth volume ratio CBCT age to be correlated with chronological age | Through study completion, an average of 1 year
  Pulp/ tooth volume ratio CBCT age to be correlated with chronological age using volumetric segmentation of CBCT software in mm3.

SECONDARY OUTCOMES:
Analysis of pulp size using linear measurements. | Through study completion, an average of 1 year
  Analysis of pulp size using linear measurements tool of CBCT software in mm.

CONTACTS AND LOCATIONS:
Overall Officials: Christine Beshara, Principal Investigator — Cairo University
Locations (1):
- Faculty of Dentistry, Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Asif MK, Nambiar P, Mani SA, Ibrahim NB, Khan IM, Lokman NB. Dental age estimation in Malaysian adults based on volumetric analysis of pulp/tooth ratio using CBCT data. Leg Med (Tokyo). 2019 Feb;36:50-58. doi: 10.1016/j.legalmed.2018.10.005. Epub 2018 Oct 21. PMID 30415192